CLINICAL TRIAL: NCT02481687
Title: The Value of Virtual Chromoendoscopy With i-SCAN and Confocal Laser Endomicroscopy in the Assessement of Dysplasia on Patients With Inflammatory Bowel Disease
Brief Title: The Value of I-Scan and Confocal Laser Endomicroscopy for the Assessment of Chronic Inflammatory Bowel Disease
Acronym: I-Scan-CLE-IBD
Status: Terminated | Type: Observational
Sponsor: University of Medicine and Pharmacy Craiova (Other)
Collaborators: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Other Study IDs: I-Scan-CLE-IBD
Record Dates: First submitted 2015-06-23; First posted 2015-06-25 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis; Dysplasia
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — One ml of whole blood and tissue biopsies from normal tissue and from modified areas of 2 to 3 mm each for molecular analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Ulcerative colitis: Consecutively admitted patients with active ulcerative colitis, confirmed by histopathology.
  I-SCAN and pCLE will be applied in all patients.
  Interventions: Other: Confocal laser endomicroscopy
- Crohn's disease: Consecutively admitted patients with active Crohn's disease, confirmed by histopathology.
  I-SCAN and pCLE will be applied in all patients.
  Interventions: Other: Confocal laser endomicroscopy

INTERVENTIONS:
Other: Confocal laser endomicroscopy — Probe based confocal laser endomicroscopy is a contrast based technique, consisting of a flexible catheter probe representing a bundle of optical fibers linked to a micro-objective a laser scanning unit and the control and acquisition software. The flexible confocal miniprobes can be passed through the working channels of standard endoscopes. The principle of the technique is based on a laser beam of defined wavelength being focused towards the targeted tissue and the recaptured signal is displayed as 'optical biopsies' in a single horizontal plane. The device was intended to be used for faster diagnosis and evaluation of gut diseases, by allowin in vivo histology.

SUMMARY:
Recently, Confocal Laser Endomicroscopy (CLE) has been developed as a novel technique that actually enables in vivo microscopic analysis of the gastrointestinal tract, during ongoing endoscopy. The potential role of CLE has been explored in pathology of both upper and lower gastrointestinal tract, showing good accuracy for predicting the final histopathological diagnosis, based on immediate evaluation of tissue and vascular patterns. Because of its minute scanning area, this techology is best used in conjunction with other "red-flag" techniques to screen the mucosa for areas of interest, which can then be examined by CLE for a histological diagnosis. I-scan technology (Pentax, Tokyo, Japan) is a new image-enhanced endoscopic technique that can achieve a virtual chromoendoscopy, but until now there have been no studies to determine the role of this technology in the evaluation of activity in inflammatory bowel disease. The study protocol is based on comparing imaging findings of p-CLE in conjunction with I-scan endoscopy with activity score and histological diagnosis of inflammatory bowel disease. CLE might have an important role in IBD patients management, by assessing the inflammation, dysplasia or response to treatment.

DETAILED DESCRIPTION:
The value of I-Scan and Confocal Laser Endomicroscopy for the assessment of chronic inflammatory bowel disease

Background Colonoscopy plays an important role in the diagnosis, assessment of activity, extension and response to therapy in chronic inflammatory bowel disease (IBD). Conventional examination underestimates extent and activity of the disease compared with histology, therefore, mucosal biopsy is a critical component of endoscopic examination of these patients. Taking multiple biopsies is time consuming, carries a low but not negligible risk of secondary hemorrahage, and causes a delay in diagnosis, whilst awaiting histological analysis.

Confocal laser endomicroscopy has emerged in recent years as a novel technique that actually enables in vivo microscopic analysis during ongoing endoscopy. Endomicroscopy can be performed either with a dedicated endoscope (eCLE) or with miniprobe-based systems (pCLE) [1]. It is a contrast based technique, the most widely used agent being the intravenously administered fluorescein [2]. The probe-based endomicroscopy system consists of a flexible catheter probe representing a bundle of optical fibers linked to a micro-objective, a laser scanning unit and the control and acquisition software (Cellvizio; Mauna Kea Technology, Paris, France). The flexible confocal miniprobes were specifically designed to be passed through the working channels of standard endoscopes, biliary catheters or cholangioscopes and thus the pCLE system can be easily integrated into any endoscopy unit. The principle of the technique is based on a laser beam of defined wavelength being focused towards the targeted tissue and the recaptured signal is displayed as 'optical biopsies' in a single horizontal plane.

The potential role of CLE has been explored in pathology of both upper and lower gastrointestinal tract, showing good accuracy for predicting the final histopathological diagnosis based on immediate evaluation of tissue and vascular patterns [3]. Because of its minute scanning area, this techology is best used in conjunction with other "red-flag" techniques to screen the mucosa for areas of interest, which can then be examined by CLE for a histological diagnosis [4].

I-scan technology (Pentax, Tokyo, Japan) is a new image-enhanced endoscopic technique, consisting of three types of algorithms: surface enhancement (SE; enhancement of the structure through recognition of the edges), contrast enhancement (CE; enhancement of depressed areas and differences in structure through colored presentation of low density areas) and tone enhancement (TE; enhancement tailored to individual organs through modification of the combination of RGB components for each pixel) [5,6]. Like narrow band imaging i-scan can achieve a virtual chromoendoscopy, but until now there have been no studies to determine the role of this technology in the evaluation of activity in inflammatory bowel disease [7].

Aim of the study The aim of the study is to compare imaging findings of p-CLE in conjunction with I-scan endoscopy with activity score and histological diagnosis.

Patients and methods The study will prospectively include patients with active ulcerative colitis or Crohn's disease who meet the inclusion and exclusion criteria. All patients will be examined by conventional colonoscopy, followed by I-scan examination and p-CLE, and biopsy samples will be taken for each segment of the colon. Then, the correlation between histology as "gold standard", activity score (Mayo score for ulcerative colitis, respectively Crohn's Disease Activity Index for Crohn's disease) and imaging findings will be calculated for both pathological and normal areas.

Inclusion criteria

* Age > 18 years old, male or female
* Patients diagnosed with active ulcerative colitis (MAYO score >3) or Crohn's disease (CDAI score >150), where an indication for treatment and colonoscopy exists. Newly diagnosed as well as patients already on oral 5-ASA therapy, may be included.
* Signed informed consent for colonoscopy and p-CLE examination Exclusion criteria
* Failure to provide informed consent
* Patients with a contraindication to colonoscopy
* Known allergy to fluorescein
* Pregnant or breast-feeding patients
* Ongoing systemic immunosuppressive therapy with prednisolone, azathioprine or biological agents.

Data collected for each participant will include:

* Personal data (name, surname, age, sex)
* Results from previous investigations
* Clinical evaluation (stools frequency, rectal bleeding, fever, abdominal pain, extra intestinal manifestation, abdominal mass) and blood count for activity index calculator (Mayo score for ulcerative colitis, respectively CDAI score for Crohn disease)
* Endoscopic findings
* Histological and immunohistochemical findings
* Molecular analysis findings

Imaging tests

* All patients will be examined by I-scan colonoscopy and the degree and distribution of the acute inflammation will be assessed.
* p-CLE examination will follow, after the intravenous administration of the contrast agent (2.5 ml fluorescein 10%), in every segment of the colon in both normal and pathological areas.
* Image data will be stored digitally for offline analysis (10-20 seconds movie for each area examined).
* Biopsy samples will be taken from each area examined by p-CLE for histological, immunohistochemical and molecular analysis.

The biological material collected during the study (this will include one ml of whole blood and tissue biopsies from normal tissue and from modified areas of 2 to 3 mm each) will be frozen and stored. When the expected number of participants is reached the samples will undergo molecular studies for assessing the markers of angiogenesis as detailed further in the protocol. The biological materials will be stored and analyzed during an estimated time of 18 months from the start of the trial. After completion of the study the biomaterials will be disposed of.

Biological samples for molecular tests:

* Blood samples will be collected before imaging procedures

  1. For DNA extraction 2-5 ml of blood can be collected in tubs containing EDTA and stored at 4°C for a day or transferred to -80°C freezer for longer storage
  2. For RNA extraction 2-5 ml of blood must be collected in PAX tubs and kept maximum 2 hours at room temperature and then transferred to -80°C freezer for longer storage
* Tissue samples:

Possible methods to stabilize tissue samples for further molecular analysis (RNA/DNA/protein):

1. 0,3-0,5 cm of tissue is stored immediately in a tube containing RNAlater Solution for approximately 24 hours at 4°C; after this the RNAlater solution is taken out from the tube (under sterile conditions) and the sample is frozen at -80°C until RNA/DNA extraction.
2. 0,3-0,5 cm of tissue is stored immediately in an empty cryogenic tube and thrown in a container that contains liquid nitrogen or dry ice with methanol.

Primary Outcome Measures:

* p-CLE findings are recorded and compared with the findings of conventional colonoscopy and I-scan colonoscopy.
* p-CLE and I-scan colonoscopy findings are compared with the pathological evaluation of tissue samples.

Secondary Outcome Measures:

* Effect of therapy, based on the results of the conventional colonoscopy, I-scan and p-CLE
* Registering time of the procedure.
* Registering possible complications

Risks and side effects Complications may occur during colonoscopy, but they are rare. These consist of bleeding at the biopsy site which is usually minimal, self-limited and rarely requires follow-up. Perforation of the bowel is extremely rare. The safety profile of the contrast agent (fluorescein) showed a very low incidence of side effects. It is not nephrotoxic and the incidence of hypersensitivity or severe allergic events is low. Fluorescein is approved for clinical use in EU countries.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old, male or female
* Patients diagnosed with active ulcerative colitis (MAYO score >3) or Crohn's disease (CDAI score >150), where an indication for treatment and colonoscopy exists. Newly diagnosed as well as patients already on oral 5-ASA therapy, may be included.
* Signed informed consent for colonoscopy and p-CLE examination

Exclusion Criteria:

* Failure to provide informed consent
* Patients with a contraindication to colonoscopy
* Known allergy to fluorescein
* Pregnant or breast-feeding patients
* Ongoing systemic immunosuppressive therapy with prednisolone, azathioprine or biological agents.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with active ulcerative colitis or Crohn's disease who meet the inclusion and exclusion criteria will be included in the study. Personal data (name, surname, age, sex), results from previous investigations, clinical evaluation (stools frequency, rectal bleeding, fever, abdominal pain, extra intestinal manifestation, abdominal mass) and blood count for activity index calculator (Mayo score for ulcerative colitis, respectively CDAI score for Crohn disease), endoscopic findings, histological and immunohistochemical findings, molecular analysis findings, will be registered in the study. p-CLE has shown its utility in both upper and lower GI tract. I-SCAN isn't widely used, so more studies are needed to prove its utility. Anyway, signed informed consent for colonoscopy, i-SCAN colonoscopy and pCLE examination is required for participation in the study
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-06; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
p-CLE findings during conventional colonoscopy and I-scan colonoscopy. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Saftoiu, MD PhD FASGE, Principal Investigator — University of Medicine and Pharmacy Craiova
Locations (1):
- Research Center of Gastroenterology and Hepatology, Craiova, Romania